CLINICAL TRIAL: NCT06458868
Title: An Open-label Controlled Trial: Effectiveness of Saltwater-UVA, Tap Water-UVA, and Bath PUVA in the Treatment of Palmoplantar Psoriasis and Contact Dermatitis.
Brief Title: An Open-label Controlled Trial: Effectiveness of Balneotherapy in Palmoplantar Psoriasis and Contact Dermatitis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hilayda Karakok Kısla, Doctor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BALNEOTERAPİ
Record Dates: First submitted 2024-05-29; First posted 2024-06-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Psoriasis; Contact Dermatitis of Hand
Keywords: bath puva; uva; psorolene; phototherapy; local uv a
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: Prospective single center open label three parallel group, adaptive randomized controlled trial
Masking Description: Endpoint assessors blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- bath puva (No Intervention): Patients received the standard protocol of bath PUVA with standard psoralen plus tap water in combination with a phototherapy regimen.
- salt water uva (Experimental): Patients received saline solution (3% NaCl) in addition to UVA with standard phototherapy regimen.
  Interventions: Other: salt water or tap water before UVA
- tap water uva (Experimental): Patients received tap water in addition to UVA with standard phototherapy regimen.
  Interventions: Other: salt water or tap water before UVA

INTERVENTIONS:
Other: salt water or tap water before UVA — Instead of using standard bath PUVA, this study investigates the efficacy of tap water or salt water with UVA in the treatment of palmoplantar psoriasis.
  Arms: salt water uva; tap water uva

SUMMARY:
Patients who had an indication for phototherapy were included in this study. The treatment was used as a monotherapy protocol.

The standard protocol for bathing PUVA involved applying 0.01% bath psoralen for 15 minutes, while the tap water group only received a tap water bath for 15 minutes and the salt water group received 3% salted (NaCl) water before UVA treatment.

Main tools to assess the efficacy is disease activity scores and quaity of Life scores.

DETAILED DESCRIPTION:
Patients who met the criteria for phototherapy were included in this study. The treatment was used as a standalone protocol, with only moisturizer permitted. In order to participate, patients needed to have completed their last systemic treatment at least 2 months prior to the study, and their last topical treatment at least 4 weeks prior.

Patients were randomized using a computer program and assessed at the beginning of therapy, as well as after 12, 24, and 36 sessions. The standard bath-PUVA protocol involved applying 0.01% bath psoralen for 15 minutes, while the tap water group only received a tap water bath for 15 minutes, and the salt water group received a 3% salt water bath before UVA exposure.

All patients were educated about their condition and current treatment options. Patients who participated in this study either had contraindications to other therapies or had experienced side effects previously.

The initial UVA dosage was 0.25 J/cm2, gradually increasing to a maximum of 5 J/cm2. During each evaluation, patients were assessed using various scales and tools to measure the severity of their psoriasis and their quality of life, as well as photographs.

Following a pilot study involving 5 patients in each group, a two score reduction in the disease activity score revealed that G power analysis determined that a total of at least 13 patients was needed to achieve 80% power. Ethical approval was obtained before commencing the study.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged between 18 and 65
* Clinical diagnosis of Palmoplantar Psoriasis or Contact Dermatitis

Exclusion Criteria:

* Individuals under 18 or over 65
* Pregnancy or breastfeeding
* History of malignancy
* Diagnosis of photodermatosis
* Prescription or use of photoallergenic or phototoxic drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2014-06-01 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Disease Severity Reduction | Disease Severity
  At least %50 reduction of the disease severity with the intervention groups at 36th week of the treatment

SECONDARY OUTCOMES:
Improvevement in the Quality of Life | Qol
  statistically significant improvement in the quality of life of the patients compared to the beginning of the study at the 36the week of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Nihal Kundakcı, Prof, Study Director — Ankara University Faculty of Medicine, Department of Dermatology and Venereology
Locations (1):
- Ankara University School of Medicine, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
If needed, a masked individual participant data is and will be stored in the archives for a duration of 5 years